CLINICAL TRIAL: NCT06758934
Title: Comparison of Textbook Outcomes Between Laparoscopic and Open Total Gastrectomy for Gastric Cancer
Status: Completed | Type: Observational
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Turgut Donmez, Ass. Prof. Dr., Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Other Study IDs: 20240213
Record Dates: First submitted 2024-12-16; First posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-12

CONDITIONS: Gastrectomy; Gastric Cancer
Keywords: Total Gastrectomy; Textbook Outcome; Open Gastrectomy; Minimally Invasive Surgery
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Open Group: Gastric cancer patients underwent open total gastrectomy with curative intent between July 2018 and January 2024
- Lap Group: Gastric cancer patients underwent laparoscopic total gastrectomy with curative intent between July 2018 and January 2024

SUMMARY:
Gastric cancer patients underwent total gastrectomy with curative intent between in a single center were included in this retrospective study. Patients divided to two groups as open and laparoscopic groups and compared in terms of demographic data, tumor characteristics, operative data and textbook outcome

DETAILED DESCRIPTION:
Gastric cancer patients underwent total gastrectomy with curative intent between July 2018 and January 2024 in a single center were included in this retrospective observational study. Enrolled patients divided to two groups as open total gastrectomy (open group) and laparoscopic total gastrectomy (lap group).

Data of patients obtained via the hospital software system. Demographic data, body mass index(BMI), Charlson comorbidity index (CCI) score and baseline characteristics, operative and postoperative results, tumor characteristics and textbook outcome results were investigated. Postoperative complications were pancreatic fistula, pleural effusion, pneumonia, anastomotic leak, intraabdominal abscess, surgical site infection, postoperative ileus.

All patients were already curative surgery patients and underwent total gastrectomy and D2 lymphadenectomy. Apart from this, the list of criteria for a patient who had a textbook outcome was as follows: no intraoperative complication, achievement of tumor-negative margins, including ≥15 harvested lymph nodes in resected specimen, no severe postoperative complication(Clavien-Dindo Score≥3, (CD)), no reintervention, no readmission to intensive care unit after once coming to the surgical ward, no prolonged hospital stay (≤21 days), no postoperative mortality (30 days) and no readmission after discharge from the hospital

ELIGIBILITY:
Inclusion Criteria:

* Gastric cancer patients underwent total gastrectomy with curative intent

Exclusion Criteria:

* Emergency surgery,
* Recurrent disease
* Metastatic disease,
* Conversion to open surgery,
* Robotic gastrectomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Gastric cancer patients ≥ 18 years old and underwent total gastrectomy with curative intent
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Textbook Outcome | 30 days
  The criteria required for a patient who underwent total gastrectomy to have reached a textbook outcome are as follows:
  * no intraoperative complication,
  * achievement of tumor-negative margin,
  * including ≥15 harvested lymph nodes in resected specimen,
  * no severe postoperative complication(Clavien-Dindo Score≥3, (CD)),
  * no reintervention,
  * no readmission to intensive care unit after once coming to the surgical ward,
  * no prolonged hospital stay (≤21 days),
  * no postoperative mortality (30 days) and
  * no readmission after discharge from the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Alpen Yahya Gümüşoğlu, Ass. Prof. Dr., Study Chair — University of Health Sciences, Bakirkoy Dr. Sadi Konuk Training and Research Hospital
Locations (1):
- Bakirkoy Dr. Sadi Konuk Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The datasets generated and analysed during the current study are not available due to institutional policies but are available from the corresponding author on reasonable request